CLINICAL TRIAL: NCT01983423
Title: Effect of Endometrial Biopsy on in Vitro Fertilization Pregnancy Rates - a Randomized, Multicenter Study
Brief Title: Effect of Endometrial Biopsy on in Vitro Fertilization Pregnancy Rates - a Multicenter Study
Acronym: EndoBx-IVF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suboptimal subject recruitment
Sponsor: Jon Havelock (Network)
Responsible Party: Sponsor-Investigator, Jon Havelock, Principal investigator, Pacific Centre for Reproductive Medicine
Organization: Pacific Centre for Reproductive Medicine (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EndoBx- IVF
Record Dates: First submitted 2013-04-12; First posted 2013-11-14 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Infertility; Pregnancy
Keywords: Endometrial Biopsy; Endometrial Sampling; In Vitro Fertilization; Pregnancy; Implantation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrial Biopsy (Experimental): Endometrial biopsy performed within 5-10 days prior to starting controlled ovarian stimulation, as part of in vitro fertilization treatment.
  Interventions: Device: Endometrial Biopsy
- Without Biopsy (No Intervention): Those proceeding with in vitro fertilization routinely, without an endometrial biopsy.

INTERVENTIONS:
Device: Endometrial Biopsy — An endometrial biopsy is performed using a sampling device known as a pipelle catheter which is introduced into the uterine cavity. The inner core is withdrawn creating suctional pressure into the hollow bore of the cavity, which allows acquisition of endometrial tissue upon rotation in the cavity. This is removed and the tissue sent for pathologic examination.
  Other Names: Endometrial pipelle biopsy; Endometrial sampling
  Arms: Endometrial Biopsy

SUMMARY:
Animal and clinical studies have suggested that local tissue trauma can promote the process of an embryo implanting in the uterine cavity. The clinical studies have been performed in patients with a history of previously failed treatments using in vitro fertilization; a process of stimulating many eggs from a women and removing them from the body, to allow fertilisation with sperm to occur in a laboratory setting. The embryos are then replaced into the uterine cavity.

This study questions whether endometrial biopsy (placing a small straw like catheter through the cervix and into the uterine cavity to take a sample of tissue via suction into the bore of the catheter), within 5-10 days of starting a cycle of in vitro fertilization, will improve pregnancy outcome for patients in the first or second cycle of treatment. The hypothesis is that endometrial biopsy will improve pregnancy outcome.

The study is a randomized multicentre study involving 3 Canadian fertility centres.

DETAILED DESCRIPTION:
Although the data are preliminary, there are studies suggesting that mild endometrial trauma in the cycle preceding IVF increases pregnancy rates, at least in women with recurrent implantation failure. Whether endometrial biopsy could promote implantation and improve pregnancy rates in the larger population of women undergoing IVF has yet to be explored. The present study will address this question and examine the impact of endometrial biopsies on IVF outcomes in the context of a randomized controlled trial.

The optimal timing of the endometrial biopsy in the cycle preceding IVF has not been determined, but the majority of the studies have included a biopsy in the mid-luteal phase of the preceding cycle. In order to allow an adjuvant therapy to IVF that would be considered tolerable to a subject, and applicable to a large infertile women population, it was determined that a single endometrial biopsy, performed approximately 1 week prior to the start of controlled ovarian hyperstimulation (COH) in an IVF cycle, would be the simplest, most flexible, and generalizable intervention to study its effects on pregnancy rates. All other components of the IVF treatment will remain constant with approximately 8-12 days of ovarian stimulation, human chorionic gonadotrophin (HCG) trigger being administered in that time frame and oocyte retrieval occuring 36 hours later from trigger. The embryo transfer will take place either day 3 or day 5 after oocyte retrieval.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing first or second IVF cycle, with or without ICSI

* Age 18-39
* BMI 18-35 kg/m2
* Uterine cavity evaluation (hysterosalpingogram, sonohysterogram, hysteroscopy) in the preceding 24 months
* Early follicular phase (Day 2 or Day 3) serum FSH, evaluated in the preceding 6 months

ONE of the following:

* Non- oral contraceptive pill (non-OCP) subjects: Documented LH surge 9-11 days prior to enrollment
* Current OCP subjects: OCP use for ≥ 10 days
* Use of long GnRH agonist or GnRH antagonist protocol
* Subject able to give informed consent

Exclusion Criteria:

* Prior enrolment in this study
* Any prior early follicular phase serum FSH level ≥12 IU/L
* Previous poor ovarian response, defined as prior IVF cycle cancelled for poor response, or ≤4 oocytes retrieved
* IVF for pre-implantation genetic diagnosis (PGD) or fertility preservation
* Diabetes mellitus or uncontrolled thyroid disease
* Abnormal uterine cavity, such as unresected submucosal fibroids, uterine septum, Mullerian anomaly such as bicornuate or unicornuate uterus or intrauterine adhesions
* Hydrosalpinx that has not been removed or surgically ligated
* Any contraindication to endometrial biopsy
* Office hysteroscopy or other uterine procedure planned or performed during cycle preceding IVF stimulation
* Use of surgically retrieved sperm

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | Five weeks gestation, as dated from the egg retrieval
  Clinical pregnancy rate, defined as transvaginal ultrasound documentation of fetal heartbeat at five weeks gestation.

SECONDARY OUTCOMES:
Implantation Rate | Five weeks gestation, as dated from the egg retrieval
  The number of gestational sacs seen at ultrasound, divided by the total number of embryos transferred
Live Birth Delivery Rate | Within twelve months of the cycle start date
  Live birth delivery rate will be the number of live birth deliveries expressed per 100 initiated cycles, aspiration cycles or embryo transfer cycles, for which the denominator (initiated, aspirated or embryo transfer cycles) will be specified. Live birth delivery will include deliveries that resulted in at least one live birth. The delivery of a singleton, twin or other multiple births will be registered as one delivery.
Fertilization Rate | 24 hours after egg retrieval
  Fertilization rate will be the number of zygotes resulting from insemination by IVF or injection by intracytoplasmic sperm injection, expressed as a ratio to the total number of oocytes inseminated or injected.
Normal Fertilization Rate | 24 Hours from egg retrieval
  Normal fertilization rate will be the number of normal zygotes resulting from insemination by IVF or injection by ICSI, expressed as a ratio to the total number of oocytes inseminated or injected.
Endometrial Thickness | Day of administration of human chorionic gonadotropin (8-12 days into ovarian stimulation)
  As assessed by transvaginal ultrasound, the maximum dimension of the endometrial cavity echo in an antero-posterior plane.
Endometrial Pattern | Day of administration of human chorionic gonadotropin (8-12 days into ovarian stimulation)
  The endometrial pattern will be categorised as either trilaminar (triple stipe pattern) or hyperechoic (diffusely echogenic)at the time of transvaginal ultrasound assessment.
Percentage of subjects with embryos cryopreserved | At the latest, day 6 after egg retrieval
  Total number of participants with embryos in excess, that met criteria for cryopreservation
The number of embryos cryopreserved per subject | At the latest, day 6 after egg retrieval
  The number of embryos each individual participant had in excess, meeting criteria for cryopreservation

CONTACTS AND LOCATIONS:
Overall Officials: Jon C Havelock, MD, Principal Investigator — Pacific Centre for Reproductive Medicine and University of British Columbia
Locations (2):
- Canada (2):
  - Pacific Centre for Reproductive Medicine, Vancouver, British Columbia
  - Mt. Sinai Hospital Centre for Fertility and Reproductive Health, Toronto, Ontario

REFERENCES:
- [Background] Lejeune B, Lecocq R, Lamy F, Leroy F. Changes in the pattern of endometrial protein synthesis during decidualization in the rat. J Reprod Fertil. 1982 Nov;66(2):519-23. doi: 10.1530/jrf.0.0660519. PMID 7175806
- [Background] Humphrey KW. The effects of some anti-oestrogens on the deciduoma reaction and delayed implantation in the mouse. J Reprod Fertil. 1968 Jul;16(2):201-9. doi: 10.1530/jrf.0.0160201. No abstract available. PMID 4298258
- [Background] Gnainsky Y, Granot I, Aldo PB, Barash A, Or Y, Schechtman E, Mor G, Dekel N. Local injury of the endometrium induces an inflammatory response that promotes successful implantation. Fertil Steril. 2010 Nov;94(6):2030-6. doi: 10.1016/j.fertnstert.2010.02.022. Epub 2010 Mar 24. PMID 20338560
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Background] Raziel A, Schachter M, Strassburger D, Bern O, Ron-El R, Friedler S. Favorable influence of local injury to the endometrium in intracytoplasmic sperm injection patients with high-order implantation failure. Fertil Steril. 2007 Jan;87(1):198-201. doi: 10.1016/j.fertnstert.2006.05.062. PMID 17197286
- [Background] Karimzadeh MA, Ayazi Rozbahani M, Tabibnejad N. Endometrial local injury improves the pregnancy rate among recurrent implantation failure patients undergoing in vitro fertilisation/intra cytoplasmic sperm injection: a randomised clinical trial. Aust N Z J Obstet Gynaecol. 2009 Dec;49(6):677-80. doi: 10.1111/j.1479-828X.2009.01076.x. PMID 20070722
- [Background] Zhou L, Li R, Wang R, Huang HX, Zhong K. Local injury to the endometrium in controlled ovarian hyperstimulation cycles improves implantation rates. Fertil Steril. 2008 May;89(5):1166-1176. doi: 10.1016/j.fertnstert.2007.05.064. Epub 2007 Aug 6. PMID 17681303
- [Background] Karimzade MA, Oskouian H, Ahmadi S, Oskouian L. Local injury to the endometrium on the day of oocyte retrieval has a negative impact on implantation in assisted reproductive cycles: a randomized controlled trial. Arch Gynecol Obstet. 2010 Mar;281(3):499-503. doi: 10.1007/s00404-009-1166-1. Epub 2009 Jul 1. PMID 19568761
- [Background] Katz VL. Diagnostic procedures. Imaging, endometrial sampling, endoscopy: indications and contraindications, complications. In: Katz VL, Lentz GM, Lobo RA, Gershenson DM, eds. Comprehensive Gynecology . 5th ed. Philadelphia, Pa: Mosby; 2007.
- [Derived] Hilton J, Liu KE, Laskin CA, Havelock J. Effect of endometrial injury on in vitro fertilization pregnancy rates: a randomized, multicentre study. Arch Gynecol Obstet. 2019 Apr;299(4):1159-1164. doi: 10.1007/s00404-019-05044-9. Epub 2019 Jan 19. PMID 30661093